CLINICAL TRIAL: NCT07217912
Title: Randomized, Double-blind Trial of Daridorexant to Prevent Delirium After Heart Surgery
Brief Title: Daridorexant to Prevent Post-cardiotomy Delirium
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Mark Oldham, Associate Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY000010860
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Cognitive Decline; Postoperative Delirium
Keywords: delirium; sleep; cognitive decline; Alzheimer disease and related dementias
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium; Delirium; Cognitive Dysfunction; Alzheimer Disease | interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio, stratified by surgery type (SAVR vs CABG) in blocks of 4, to receive either daridorexant or matching placebo on the first three postoperative nights following heart surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug and placebo will be identical in appearance, labeling, and administration schedule. Randomization and treatment assignment will be managed by the investigational pharmacy. The blind will be maintained for participants, care providers, investigators, and outcome assessors, and will be broken only after data lock or in the event of a medical emergency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- daridorexant (Experimental): Oral daridorexant 50 mg (or 25 mg, if taking a moderate 3A4 inhibitor) each of the first three nights after heart surgery.
  Interventions: Drug: Daridorexant 50 mg
- placebo (Placebo Comparator): Oral matching placebo each of the first three nights after heart surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Daridorexant 50 mg — Administered consistent with labeling from the US Food and Drug Administration.
  Arms: daridorexant
Other: Placebo — Identical appearing to daridorexant
  Arms: placebo

SUMMARY:
The goal of this follow-on pilot randomized clinical trial is to obtain additional preliminary data to inform a larger, adequately powered phase 2b trial of daridorexant for the prevention of postoperative delirium after heart surgery. Having demonstrated feasibility in a prior study (RSRB #9841), this study aims to estimate the effect of daridorexant on (1) reducing delirium symptom burden and incidence and (2) improving self-reported sleep quality during the postoperative period, and (3) to assess the feasibility of collecting objective sleep data in the postoperative setting.

Participants will: complete a baseline visit; take the study drug, either daridorexant or placebo, each of the first three nights after heart surgery; and be evaluated daily for sleep and delirium during the first three postoperative days. Participants will also have the option of wearing a sleep monitor in the hospital each of the first three nights after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 yrs;
* having surgical aortic valve surgery or coronary artery bypass graft surgery at Strong Memorial Hospital;
* can provide consent;
* able to speak, read,and write English (as the instruments, including semi-structured interviews, used in this protocol have been validated in English);
* family member or close friend for collateral.

Exclusion Criteria:

* Prior cardiotomy
* Infectious endocarditis
* Emergency surgery
* Delirium at baseline (positive 3D-CAM)
* Auditory or visual impairment that prevents study procedures
* Alcohol or substance misuse (CAGE-AID score ≥ 2)
* Psychotic disorder
* Dementia-level deficits (TICS < 27)
* Use of a prescription sleep aid at least every other night
* Use of a strong CYP3A4 inhibitor (e.g., ceritinib, clarithromycin, cobicistat, idelalisib, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, telithromycin, voriconazole)
* Daridorexant intolerance
* Severe kidney or liver impairment (Child-Pugh ≥7, Cockcroft-Gault <30 mL/min, or on dialysis)
* Narcolepsy
* Suicidal ideation at baseline
* Any condition that, in the PI's opinion, compromises patient safety or data quality
* Additional exclusions for the NLP exploratory aim: history of traumatic brain injury or head concussions with loss of consciousness, use of corticosteroids, or history of major neurological disease or brain surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Delirium incidence and severity | Postoperative Days 1-3
  Participants will be assessed on postoperative days 1-3 using the Delirium Rating Scale, Revised-98 (DRS-R98; range 0-39; higher scores indicate greater severity of delirium symptoms) and 3-minute Diagnostic interview for the Confusion Assessment Method (3D-CAM; 22 dichotomous items used to inform delirium status). Delirium diagnosis is defined per Diagnostic and Manual of Mental Disorders, 5th Edition, Text Revision, and its severity defined as the sum of DRS-R98 score on postoperative days 1-3.

SECONDARY OUTCOMES:
Postoperative sleep quality | Postoperative Nights 1-3
  Participants will complete Richards-Campbell Sleep Questionnaire on postoperative days 1-3. This scale includes 6 items (sleep-related domains), each scored using a visual analog scale, ranging from 0 to 100. The total score represents the mean of the first five domain scores. Higher scores indicate better subjective sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No